CLINICAL TRIAL: NCT06216210
Title: Assessing the Impact of Opioid-Free Anesthesia Using the Modified Mulimix Technique on Plasma Interleukin-2 and Interleukin-6 Levels in Bariatric Surgery Patients
Brief Title: Assessing the Impact of Opioid-Free Anesthesia Using the Modified Mulimix Technique.
Acronym: Mulimi
Status: Completed | Type: Observational
Sponsor: Zulekha Hospitals (Other)
Responsible Party: Sponsor
Other Study IDs: T.G.H.45/275
Record Dates: First submitted 2023-12-26; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Opioid Use

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group (A): Opioid-free anesthesia group
  Interventions: Drug: opioid-FREE anesthesia.
- Group (B): Opioid-containing anesthesia group.
  Interventions: Drug: opioid-CONTAINING anesthesia.

INTERVENTIONS:
Drug: opioid-FREE anesthesia. — They received opioid-free anesthesia. These patients were provided a multimodal combination infusion. The administration of this infusion commenced at a dosage of 0.2 micrograms per kilogram per hour of dexmedetomidine. The "Modified Mulimix" cocktail, consisting of dexmedetomidine at a concentration of 10 ug/ml, Ketamine at a concentration of 2.5 mg/ml, and Lignocaine at a concentration of 20 mg/ml, was administered to a patient weighing 100 kg and if the weight is 110 Kg the rate will be increased by 10 percent, etc.,
  Other Names: GROUP (A)
  Groups: Group (A)
Drug: opioid-CONTAINING anesthesia. — The process of inducing anesthesia included the injection of fentanyl at a dosage of 2 micrograms per kilogram during the induction phase. Additionally, morphine was administered at a dose of 0.03 milligrams per kilogram at the time of port insertion.
  Other Names: GROUP (B)
  Groups: Group (B)

SUMMARY:
The effective management of post-operative pain in the setting of bariatric surgery presents significant hurdles for both anesthesiologists and surgeons. The objective of this study was to assess the effects of opioid-free anesthesia (OFA) using the modified mulimix technique on the levels of plasma interleukin-2 (IL-2) and interleukin-6 (IL-6) as the primary outcome. Additionally, the study aimed to evaluate the duration of analgesia and the analgesic requirements within the first twenty-four hours after surgery.

DETAILED DESCRIPTION:
Objectives: The effective management of post-operative pain in the setting of bariatric surgery presents significant hurdles for both anesthesiologists and surgeons. The objective of this study was to assess the effects of opioid-free anesthesia (OFA) using the modified mulimix technique on the levels of plasma interleukin-2 (IL-2) and interleukin-6 (IL-6) as the primary outcome. Additionally, the study aimed to evaluate the duration of analgesia and the analgesic requirements within the first twenty-four hours after surgery.

Methods: 60 patients were systematically selected and randomly assigned to Group A (OFA) and Group B (Opioid-Containing Anesthesia, OCA), with the modified Mulimix technique employed. Serum samples were collected from all patients, both at the onset of the skin incision and after the surgical procedure. These samples were then used to assess interleukin-2 (IL-2) and interleukin-6 (IL-6) levels. Additionally, the post-operative analgesic consumption was documented.

ELIGIBILITY:
Inclusion Criteria:

* both genders
* aged between 20 and 50 years
* patients fall under the American Society of Anesthesia (ASA) categories II-III
* body mass index (BMI) ranging from 35-50.

Exclusion Criteria:

* patients who declined participation in the trial
* pregnant women
* patients who encountered challenges in communication that could potentially impede a dependable postoperative evaluation

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A study was conducted on a sample of 60 patients, comprising individuals of both genders aged between 20 and 50 years.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2023-10-04 (Actual); Study Completion 2023-10-04 (Actual)

PRIMARY OUTCOMES:
immunological response | 20 MONTHS
  to detect the immunological response in the form of IL-2 and IL-6.

SECONDARY OUTCOMES:
The analgesic duration and requirements in the first twenty-four hours postoperatively | 20 MONTHS
  assessing the analgesic duration and requirements in the first twenty-four hours postoperatively
comparing the Visual Analog Score | 20 MONTHS
  comparing the Visual Analog Score between opioid-free anesthesia and opioid-contained. anesthesia. scale values from 0 to 100. from 0 to 4 considered no pain
The Non-Invasive blood pressure at baseline, 2 hours, 4 hours, 6 hours, 12 hours and 24 hours. | 20 MONTHS
  investigating the changes in blood pressure associated with the two different anesthetic techniques to determine the most suitable approach for bariatric surgery.
Heart rate at baseline, 2 hours, 4 hours, 6 hours, 12 hours and 24 hours. | 20 MONTHS
  investigating the changes in heart rate associated with the two different anesthetic techniques to determine the most suitable approach for bariatric surgery.

CONTACTS AND LOCATIONS:
Overall Officials: SAMEH HA SEYAM, MD, Study Chair — assistant professor of anesthesiology, intensive care, and pain management, A-Azhar university
Locations (1):
- Al-Azhar faculty of medicine, Cairo, Egypt